CLINICAL TRIAL: NCT05841732
Title: MyBack - Effectiveness and Implementation of a Behavior Change Informed Exercise Program to Prevent Low Back Pain Recurrences: a Hybrid Effectiveness-implementation Randomized Controlled Study
Brief Title: MyBack - A Behavior Change Informed Exercise Program to Prevent Low Back Pain Recurrences
Acronym: MyBack
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Setúbal (Other)
Collaborators: Universidade Nova de Lisboa (Other)
Responsible Party: Principal Investigator, Eduardo B. Cruz, Professor, Instituto Politécnico de Setúbal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PTDC/SAU-SER/7406/2020
Record Dates: First submitted 2023-04-11; First posted 2023-05-03 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain
Keywords: Low back pain; Recurrences; Exercise; Behaviour change; Primary health care
MeSH Terms: conditions — Low Back Pain; Recurrence; Motor Activity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Other): Participants allocated to the usual care group will be informed that they can access their GP in the usual way (GPs consultation, pain medication, referral for other treatments/ services) and that they should contact their GP if their condition worsens. In addition, they will receive a minimal educational intervention focused on symptom management and promotion of physical activity ("stay active").
  Interventions: Other: Usual Care
- MyBack (Experimental): Patients in the MyBack group will participate in a patient-centred, tailored exercise programme informed by a behavioural change approach in addition to receiving usual care. The MyBack intervention programme will consist of 12 bi-weekly sessions (60 minutes each) over 6 weeks complemented by 12 exercise sessions to be carried out autonomously by the participants over the following 6 weeks
  Interventions: Other: Usual Care; Other: MyBack Program

INTERVENTIONS:
Other: Usual Care — Education; Pain Medication, imaging, referrals to other health services, other health care appointments
  Other Names: Minimal intervention
Other: MyBack Program — A tailored exercise and behavioural change program
  Other Names: Physiotherapy
  Arms: MyBack

SUMMARY:
Low Back Pain is a common heath condition with high rates of recurrence and huge associated costs. Research has focused its efforts on analysing the effects of interventions while knowledge about effective secondary prevention strategies is limited. MyBack study aims to analyse the effectiveness of a tailored exercise and behavioural change program (MyBack program) in the secondary prevention of low back pain, and evaluate acceptability, feasibility and determinants of implementation by the different stakeholders, as well as the implementation strategy of the MyBack program, through a hybrid type I, randomized, controlled and multicentre study of effectiveness and implementation in the context of primary health care.

ELIGIBILITY:
Inclusion Criteria:

* Recovered (within the last 3 months) from an episode of non-specific LBP (with or without leg pain and of any duration)
* Recovery from an LBP episode is defined as having a pain score of "0" or "1" on a 11-point Numeric Pain Rating Scale for, at least, 30 consecutive days
* Age between 18 and 65 years;
* Read and speak the Portuguese language;
* Having a mobile phone capable of receiving and sending text messages;
* No medical contraindication to exercise.

Exclusion Criteria:

* Diagnosis, or symptoms consistent with, severe depression or other psychiatric condition,
* Pregnancy
* Spinal surgery in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Risk of low back pain recurrence | 1 month after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected.
Risk of low back pain recurrence | 2 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected.
Risk of low back pain recurrence | 3 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected.
Risk of low back pain recurrence | 4 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected.
Risk of low back pain recurrence | 5 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected.
Risk of low back pain recurrence | 6 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected.
Risk of low back pain recurrence | 7 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected.
Risk of low back pain recurrence | 8 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected.
Risk of low back pain recurrence | 9 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected.
Risk of low back pain recurrence | 10 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected.
Risk of low back pain recurrence | 11 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected.
Risk of low back pain recurrence | 12 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected.

SECONDARY OUTCOMES:
Pain intensity | Baseline, 3, 6 and 12 months after baseline
  Pain intensity will be measured with a 11-point Numeric Pain Rating Scale. Total scores range from 0 to 10, with higher scores indicating higher levels of pain.
Functional Disability | Baseline, 3, 6 and 12 months after baseline
  Functional Disability will be measured through the Roland Morris Disability Questionnaire (RMDQ). Total scores range from 0 to 24, with higher scores indicating higher levels of functional disability.
Musculoskeletal Health | Baseline, 3, 6 and 12 months after baseline
  Musculoskeletal Health will be measured through the Musculoskeletal Health Questionnaire (MSK-HQ). Total scores range from 0 to 56, with higher scores indicating higher levels of musculoskeletal health.
Health-related quality of life | Baseline, 3, 6 and 12 months after baseline
  Health-related Quality of life (HRQoL) will be measured by the EuroQuol 5 dimensions, 5 levels questionnaire. Total scores range from 0 to 1, with higher scores indicating higher levels of health-related quality of life.
Medical appointments for a low back pain recurrence | 3, 6, 9 and 12 months after baseline
  The number of primary care visits to the General Practitioner for a low back pain recurrence, for each participant, will be collected from the local medical records
Imaging tests prescribed related with a low back pain recurrence | 3, 6, 9 and 12 months after baseline
  The number of x-rays, MRI and CT-scans of lower back will be collected for each participant from the local medical records
Pain medication for low back pain recurrence | 3, 6, 9 and 12 months after baseline
  The number and name of the medication prescribed will be collected for each participant from the local medical records
Referral to other interventions and sickness certificates | 3, 6, 9 and 12 months after baseline
  Referral to other interventions or to other medical specialities or services or sickness certificates will be recorded will be collected for each participant from the local medical records.
Impact of LBP recurrence | 1 month after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected. In the presence of a LBP recurrence, pain intensity (11-point Numeric Pain Rating Scale), functional disability (Roland Morris Disability Questionnaire), care seeking (number of primary care visits, imaging tests prescribed and pain medication) and work status (sick leave: yes/no) will be collected by telephone.
Impact of LBP recurrence | 2 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected. In the presence of a LBP recurrence, pain intensity (11-point Numeric Pain Rating Scale), functional disability (Roland Morris Disability Questionnaire), care seeking (number of primary care visits, imaging tests prescribed and pain medication) and work status (sick leave: yes/no) will be collected by telephone.
Impact of LBP recurrence | 3 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected. In the presence of a LBP recurrence, pain intensity (11-point Numeric Pain Rating Scale), functional disability (Roland Morris Disability Questionnaire), care seeking (number of primary care visits, imaging tests prescribed and pain medication) and work status (sick leave: yes/no) will be collected by telephone.
Impact of LBP recurrence | 4 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected. In the presence of a LBP recurrence, pain intensity (11-point Numeric Pain Rating Scale), functional disability (Roland Morris Disability Questionnaire), care seeking (number of primary care visits, imaging tests prescribed and pain medication) and work status (sick leave: yes/no) will be collected by telephone.
Impact of LBP recurrence | 5 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected. In the presence of a LBP recurrence, pain intensity (11-point Numeric Pain Rating Scale), functional disability (Roland Morris Disability Questionnaire), care seeking (number of primary care visits, imaging tests prescribed and pain medication) and work status (sick leave: yes/no) will be collected by telephone.
Impact of LBP recurrence | 6 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected. In the presence of a LBP recurrence, pain intensity (11-point Numeric Pain Rating Scale), functional disability (Roland Morris Disability Questionnaire), care seeking (number of primary care visits, imaging tests prescribed and pain medication) and work status (sick leave: yes/no) will be collected by telephone.
Impact of LBP recurrence | 7 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected. In the presence of a LBP recurrence, pain intensity (11-point Numeric Pain Rating Scale), functional disability (Roland Morris Disability Questionnaire), care seeking (number of primary care visits, imaging tests prescribed and pain medication) and work status (sick leave: yes/no) will be collected by telephone.
Impact of LBP recurrence | 8 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected. In the presence of a LBP recurrence, pain intensity (11-point Numeric Pain Rating Scale), functional disability (Roland Morris Disability Questionnaire), care seeking (number of primary care visits, imaging tests prescribed and pain medication) and work status (sick leave: yes/no) will be collected by telephone.
Impact of LBP recurrence | 9 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected. In the presence of a LBP recurrence, pain intensity (11-point Numeric Pain Rating Scale), functional disability (Roland Morris Disability Questionnaire), care seeking (number of primary care visits, imaging tests prescribed and pain medication) and work status (sick leave: yes/no) will be collected by telephone.
Impact of LBP recurrence | 10 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected. In the presence of a LBP recurrence, pain intensity (11-point Numeric Pain Rating Scale), functional disability (Roland Morris Disability Questionnaire), care seeking (number of primary care visits, imaging tests prescribed and pain medication) and work status (sick leave: yes/no) will be collected by telephone.
Impact of LBP recurrence | 11 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected. In the presence of a LBP recurrence, pain intensity (11-point Numeric Pain Rating Scale), functional disability (Roland Morris Disability Questionnaire), care seeking (number of primary care visits, imaging tests prescribed and pain medication) and work status (sick leave: yes/no) will be collected by telephone.
Impact of LBP recurrence | 12 months after baseline
  Participants will receive a text message with a yes/no question regarding low back pain recurrence. The number of participants with a recurrence of low back pain, defined as the return of LBP with a minimum duration of 24 hours, with a pain intensity ≥2 on an 11-point numerical scale, preceded by a minimum period of 30 days without pain, will be collected. In the presence of a LBP recurrence, pain intensity (11-point Numeric Pain Rating Scale), functional disability (Roland Morris Disability Questionnaire), care seeking (number of primary care visits, imaging tests prescribed and pain medication) and work status (sick leave: yes/no) will be collected by telephone.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Cruz, PhD, Principal Investigator — Instituto Politécnico de Setúbal
Locations (1):
- Instituto Politécnico de Setúbal, Setúbal, Setúbal District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pires D, Duarte S, Rodrigues AM, Caeiro C, Canhao H, Branco J, Alves J, Marques M, Aguiar P, Fernandes R, Sousa RD, Cruz EB. MyBack - effectiveness and implementation of a behavior change informed exercise programme to prevent low back pain recurrences: a hybrid effectiveness-implementation randomized controlled study protocol. BMC Musculoskelet Disord. 2024 Jun 5;25(1):440. doi: 10.1186/s12891-024-07542-7. PMID 38840084